CLINICAL TRIAL: NCT02972372
Title: A Randomized, Open-label, Multicenter Trial of the Chemoradiation Versus Standard Esophagectomy for Locally Advanced Resectable Esophageal Squamous Cell Cancer in Chinese Patients
Brief Title: Chemoradiation Versus Esophagectomy for Locally Advanced Esophageal Cancer
Acronym: CELAEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry); Anyang Tumor Hospital (Other); 150th Hospital of PLA (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRTESC6111
Record Dates: First submitted 2016-11-06; First posted 2016-11-23 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Esophagus Cancer
Keywords: esophageal cancer; chemoradiation; esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Chemoradiotherapy; Surgical Procedures, Operative; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- CRT group (Active Comparator): 3-weekly cycles of cisplatin and 5-fluorouracil chemotherapy and radical radiotherapy delivered in IMRT mode (total of 50Gy given in 25 fractions) will be given over a period 5-6 weeks.
  Interventions: Procedure: CRT
- Surgery group (Active Comparator): The patients randomized to receive either standard esophagectomy will have the operation performed in an open manner with two-field lymphadenectomy
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: CRT — Drug: Capecitabine(Aibin) capecitabine(Aibin)：625mg/m2, bid d1-5; q1w, po,5 weeks in total
  Other Names:
  Aibin Drug: Oxaliplatin(Aiheng) Oxaliplatin(Aiheng)：65mg/m2，d1，8, 22, 29,I.V.
  Other Names:
  Aiheng cisplatin: 75mg/m2 d1，29 or d1, 29, 57, 85. 5-Fu：750mg/m2 CIV24h d1-4，d29-32 or d1-4，d29-32, d57-60, d85-88.
  Radiation: Radiotherapy concurrent radiotherapy：IMRT radiotherapy 50Gy in total，2 Gy/d，5d/w，Until disease progression or unacceptable toxicity
  Other Names: concurrent chemoradiotherapy
  Arms: CRT group
Procedure: surgery — The patients randomized to receive either standard esophagectomy will have the operation performed in an open manner with two-field lymphadenectomy
  Other Names: esophagectomy
  Arms: Surgery group

SUMMARY:
The aim of this study is to compare outcomes in Chinese patients with locally advanced resectable esophageal squamous cell cancer who have received either surgery or definitive chemoradiation (CRT) by the randomized, open-label, multicenter trial.

DETAILED DESCRIPTION:
Background: More than half of global esophageal cancer cases came from China, but the report about definitive chemoradiation (CRT) compared with esophagectomy in Chinese patients with locally advanced resectable esophageal squamous cell cancer (ESCC) is limited.

Aim: to compare outcomes in Chinese patients with locally advanced resectable esophageal squamous cell cancer who have received either surgery or definitive chemoradiation (CRT).

Methods: 176 ESCC patients with T1bN+M0, T2-4aN0-2M0 will be randomized to CRT group or Surgery group.In the CRT group, patients will be given intensity modulation radiation therapy (IMRT) with 50Gy/25 fractions , and current chemotherapy with 5-fluorouracil (5-FU) basic regimens. In the surgery group, patients will received standard esophagectomy. 5 years follow-up for both groups patients.

Primary endpoints: 2 year and 5 year Disease free survival, Overall survival Second endpoints: treatment-related adverse events; the quality of life

ELIGIBILITY:
Inclusion Criteria:

* Chinese
* esophageal squamous cell cancer
* mid or lower esophageal cancer
* tumor is resectable disease
* clinical stage: cT1bN+Mo, or cT2-4aN0-2M0

Exclusion Criteria:

* who had distant metastasis to solid visceral organs or local invasion into trachea, descending aorta, or recurrent laryngeal nerve.
* who had a serious premorbid condition or a poor physical status that compromised a thoracotomy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival rate | 2 year
  The percent of 2 year disease-free survival after random allocation, percent

SECONDARY OUTCOMES:
Treatment-related adverse events | 2 year
  The percent of treatment-related adverse events after 2 year random allocation, percent
QoF (quality of life) | 2 year
  The quality of life evaluation after 2 year of random allocation by questionnaire, 1-10 score, 1 means poor and 10 means best
2 year overall survival | 2 year
  The percent of 2 year overall survival after random allocation, percent

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, MD, PhD, Study Chair — The First Affiliated Hospital, and College of Clinical Medicine of Henan University of Science and Technology; Fuyou Zhou, MD, PhD, Study Chair — Anyang Tumor Hospital; Ruinuo Jia, MD, Principal Investigator — The First Affiliated Hospital, and College of Clinical Medicine of Henan University of Science and Technology
Locations (2):
- China (2):
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital, and College of Clinical Medicine of Henan University of Science and Technology, Luoyang, Henan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teoh AY, Chiu PW, Yeung WK, Liu SY, Wong SK, Ng EK. Long-term survival outcomes after definitive chemoradiation versus surgery in patients with resectable squamous carcinoma of the esophagus: results from a randomized controlled trial. Ann Oncol. 2013 Jan;24(1):165-71. doi: 10.1093/annonc/mds206. Epub 2012 Aug 10. PMID 22887465
- [Background] Teoh AY, Yan Chiu PW, Wong TC, Liu SY, Hung Wong SK, Ng EK. Functional performance and quality of life in patients with squamous esophageal carcinoma receiving surgery or chemoradiation: results from a randomized trial. Ann Surg. 2011 Jan;253(1):1-5. doi: 10.1097/SLA.0b013e3181fcd991. PMID 21233603
- [Background] Park JW, Kim JH, Choi EK, Lee SW, Yoon SM, Song SY, Lee YS, Kim SB, Park SI, Ahn SD. Prognosis of esophageal cancer patients with pathologic complete response after preoperative concurrent chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):691-7. doi: 10.1016/j.ijrobp.2010.06.041. Epub 2010 Oct 1. PMID 20888705
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Blum MA, Taketa T, Sudo K, Wadhwa R, Skinner HD, Ajani JA. Chemoradiation for esophageal cancer. Thorac Surg Clin. 2013 Nov;23(4):551-8. doi: 10.1016/j.thorsurg.2013.07.006. PMID 24199704
- [Background] Conroy T, Galais MP, Raoul JL, Bouche O, Gourgou-Bourgade S, Douillard JY, Etienne PL, Boige V, Martel-Lafay I, Michel P, Llacer-Moscardo C, Francois E, Crehange G, Abdelghani MB, Juzyna B, Bedenne L, Adenis A; Federation Francophone de Cancerologie Digestive and UNICANCER-GI Group. Definitive chemoradiotherapy with FOLFOX versus fluorouracil and cisplatin in patients with oesophageal cancer (PRODIGE5/ACCORD17): final results of a randomised, phase 2/3 trial. Lancet Oncol. 2014 Mar;15(3):305-14. doi: 10.1016/S1470-2045(14)70028-2. Epub 2014 Feb 18. PMID 24556041
- [Background] Kato K, Muro K, Minashi K, Ohtsu A, Ishikura S, Boku N, Takiuchi H, Komatsu Y, Miyata Y, Fukuda H; Gastrointestinal Oncology Study Group of the Japan Clinical Oncology Group (JCOG). Phase II study of chemoradiotherapy with 5-fluorouracil and cisplatin for Stage II-III esophageal squamous cell carcinoma: JCOG trial (JCOG 9906). Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):684-90. doi: 10.1016/j.ijrobp.2010.06.033. Epub 2010 Oct 6. PMID 20932658
- [Background] Kato K, Nakajima TE, Ito Y, Katada C, Ishiyama H, Tokunaga SY, Tanaka M, Hironaka S, Hashimoto T, Ura T, Kodaira T, Yoshimura K. Phase II study of concurrent chemoradiotherapy at the dose of 50.4 Gy with elective nodal irradiation for Stage II-III esophageal carcinoma. Jpn J Clin Oncol. 2013 Jun;43(6):608-15. doi: 10.1093/jjco/hyt048. Epub 2013 Apr 12. PMID 23585687
- [Background] Lee SJ, Ahn BM, Kim JG, Sohn SK, Chae YS, Moon JH, Lee EB, Kim JC, Park IK, Jeon SW. Definitive chemoradiotherapy with capecitabine and cisplatin in patients with esophageal cancer: a pilot study. J Korean Med Sci. 2009 Feb;24(1):120-5. doi: 10.3346/jkms.2009.24.1.120. Epub 2009 Feb 28. PMID 19270824
- [Background] Xing L, Liang Y, Zhang J, Wu P, Xu D, Liu F, Yu X, Jiang Z, Song X, Zang Q, Wang W. Definitive chemoradiotherapy with capecitabine and cisplatin for elder patients with locally advanced squamous cell esophageal cancer. J Cancer Res Clin Oncol. 2014 May;140(5):867-72. doi: 10.1007/s00432-014-1615-5. Epub 2014 Mar 1. PMID 24578238
- [Derived] Jia R, Yin W, Li S, Li R, Yang J, Shan T, Zhou D, Wang W, Wan L, Zhou F, Gao S. Chemoradiation versus oesophagectomy for locally advanced oesophageal cancer in Chinese patients: study protocol for a randomised controlled trial. Trials. 2019 Apr 11;20(1):206. doi: 10.1186/s13063-019-3316-5. PMID 30971301